CLINICAL TRIAL: NCT02490644
Title: Role of High Mobility Group Box 1 as a Prognostic Biomarker in Patients Undergoing Valvular Heart Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0764
Record Dates: First submitted 2015-06-30; First posted 2015-07-07 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MGB1 in valvular heart surgery: Evaluation of the high mobility group box 1 as a prognostic biomarker in patients undergoing valvular heart surgery
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling 5ml

SUMMARY:
One of the most important factor that affects the post op complication of the cardiac surgery is systemic inflammation. Valvular heart surgery requires cardiopulmonary bypass and cardioplegic arrest, which can arouse the ischemic/reperfusion injury causing myocardial damage and inflammatory response. These myocardial damage and inflammatory response can cause multi-organ failure or even death.

DETAILED DESCRIPTION:
One of the most important factor that affects the post op complication of the cardiac surgery is systemic inflammation. Valvular heart surgery requires cardiopulmonary bypass and cardioplegic arrest, which can arouse the ischemic/reperfusion injury causing myocardial damage and inflammatory response. These myocardial damage and inflammatory response can cause multi-organ failure or even death.

High-mobility group protein B1 (HMGB1) is a protein which is encoded by the HMGB1 gene in human. HMGB1 is secreted by immune cells (like macrophages, monocytes and dendritic cells). Activated macrophages and monocytes secrete HMGB1 as a cytokine mediator of Inflammation. There are many studies suggesting the relationship between HMGB1 and acute coronary syndrome, myocardial ischemic/reperfusion injury, atherosclerosis, heart failure and other cardiac disease as a marker for inflammatory response. However, there are no other study evaluating HMGB1 as a prognostic factor after valvular surgery, so far.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20
* patients undergoing aortic valve surgery or more than single valve surgery

Exclusion Criteria:

* age < 20
* patients undergoing single mitral valve surgery
* history of open heart surgery
* emergency surgery
* history of steroid medication
* infective disease and/or malignant tumor
* coronary artery bypass surgery or aortic replacement surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people who undergo valvular heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-01-12; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
concentration of HMGB1 | collect blood sample right before the surgery after induction of anesthesia
  The relationship between concentration of HMGB1 and post op prognosis in patients undergoing valvular heart surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea